CLINICAL TRIAL: NCT02984748
Title: Prediction of Outcomes in Adult Cochlear Implant Recipients
Brief Title: Outcome Prediction in Cochlear Implant Recipients
Status: Completed | Type: Observational
Sponsor: The Hearing Cooperative Research Centre (Other)
Collaborators: Cochlear (Industry); Attune Hearing (Unknown); Sydney Cochlear Implant Clinic (Unknown)
Responsible Party: Sponsor
Other Study IDs: CLTD 5565
Record Dates: First submitted 2016-12-04; First posted 2016-12-07 (Estimated); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Hearing Loss
Keywords: cochlear implants; hearing loss
MeSH Terms: conditions — Hearing Loss | interventions — Cochlear Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cochlear Implant Recipients
  Interventions: Device: Cochlear implant

INTERVENTIONS:
Device: Cochlear implant

SUMMARY:
The ability to predict post-operative outcomes after implantation is important for a number of reasons, including being able to advise candidates of appropriate expectations using evidence based guidance. The approved study involves investigation of the ability to predict outcomes in the implanted ear alone and in the best-aided binaural listening conditions, examining a number of measured factors both pre-, peri- and post-operatively. The study incorporates a range of functional outcome measures through questionnaires to ascertain social, functional and demographic factors that may be predictive of outcomes. Questionnaires are also administered to determine the degree of benefit obtained after implantation for each individual, since this forms a key component of providing pre-operative counselling to candidates.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical suitability for first side implantation, i.e. not undergoing assessment for second side cochlear implant surgery
2. Willing and able to attend the study visits
3. Able to provide informed consent for participation in the study, with an understanding of the requirements, risks and benefits of participation in the investigation
4. Able to read and understand study documents and follow investigator instructions
5. Able to understand and follow study personnel instructions during audiological measurements
6. Native speaker in the language used to assess clinical speech perception performance

Exclusion Criteria:

1. Unrealistic expectations on the part of the subject regarding the possible benefits, risks, and limitations that are inherent to enrolment in the clinical investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Cochlear Implant Recipients
Sampling Method: Non-Probability Sample
Enrollment: 267 (Actual)
Dates: Start 2014-10-07 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Speech recognition in quiet | Testing over 12 months
  Speech recognition scores in quiet
Speech recognition in noise | Testing over 12 months
  Speech recognition scores in noise

CONTACTS AND LOCATIONS:
Locations (1):
- The HEARing CRC, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No